CLINICAL TRIAL: NCT05203042
Title: Comparison of Cognitive and Motor Dual Task Performance in Individuals With Prediabetes and Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Gizem Mermerkaya, Lecturer, Bartın Unıversity
Other Study IDs: BartınU
Record Dates: First submitted 2021-10-02; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Prediabetes; Double task performance
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- prediabetes
- diabetes

SUMMARY:
The aim of this study is to compare the dual task task in individuals with prediabetes and diabetes. According to the results of this study, if there is a difference in dual-task performances and other conditions between people with prediabetes and people with diabetes, it will be a reference study for intervention studies accordingly.

DETAILED DESCRIPTION:
Diabetes is a chronic, broad-spectrum metabolic disorder that requires continuous medical care, in which the organism cannot adequately benefit from carbohydrates, fats and proteins due to insulin deficiency or defects in the effect of insulin. The number of diabetes cases worldwide has increased rapidly over the past four decades, rising from 108 million in 1980 to 422 million in 2014 . An aging population, physical inactivity, and rising obesity rates are recognized as driving factors for the rapid growth of diabetes . Diabetes is a leading cause of mortality and is a strong risk factor for both microvascular and macrovascular complications . Adequate glycemic control, cardiovascular risk factors management, early treatment of complications and related comorbidities are required for appropriate Type 2 Diabetes management . Complications of Type 2 Diabetes include heart and blood vessel disease, neuropathy, kidney disease, skin and eye damage, sleep apnea, bone metabolism disorders, mood disorders, and cognitive impairment. Therefore, it is essential to maintain a healthy lifestyle with weight control, balanced diet, smoking cessation, and physical activity The concept of prediabetes includes individuals who do not meet the criteria for a diagnosis of diabetes, but whose blood sugar is above normal limits. In other words, it can be called the pre-diabetic period when glucose metabolism begins to deteriorate. In a study conducted by the Centers for Disease Control and Prevention (CDC) in the United States in 2014, it was shown that there are 29 million adults with diabetes and 86 million adults with prediabetes in the United States. In another study, it was predicted that there would be more than 470 million individuals with prediabetes worldwide in 2030. Prediabetic individuals are more likely to develop diabetes than healthy individuals. Although the rate of progression varies in the literature, it has been reported that 5-10% of prediabetic individuals become diabetic every year. At the same time, many studies conducted around the world have shown that the risk of many comorbidities in diabetes and prediabetes is the same and affects all age groups. In conclusion, prediabetes is a toxic cardiometabolic condition associated with an increased risk for microvascular and macrovascular complications. Given the millions of people with prediabetes worldwide, identifying and responding to at-risk prediabetic populations is critical to contain the increased risks of cardiometabolic disease and conversion rates to diabetes.In a 10-year follow-up study conducted in prediabetes and diabetics, a linear relationship was found between individuals' HbA1c levels and cognitive decline. At the same time, evidence has shown that poor glycemic control is strongly associated with the development of cognitive dysfunction. Cerebral and peripheral vascular complications (eg, neuropathy, white matter disease, stroke, myocardial infarction, peripheral artery disease) that develop as a result of chronic exposure to hyperglycemia have been associated with cognitive impairment in Type 2 diabetes. Affected cognitive areas are reported as decreased psychomotor speed, impaired memory, executive processes, and attention. Executive processes are "higher-level" functions that monitor and control other cognitive processes. These capacities are thought to underlie activities such as planning, making decisions, switching tasks, goal-directed behavior, and coordinating ongoing activities (for example, doing two things at once or planning a series of activities). More importantly, it is critical for sensory integration used to coordinate executive function, balance, and gait motor output.Dual task paradigms are used to examine the degree of automaticity of movement. In these paradigms, a primary task is undertaken, often such as walking, which is the main focus of attention. Secondary tasks are added and the resulting impact on both tasks is examined. In everyday situations it is normal to undertake multiple tasks at once, such as walking and talking, so these situations are essentially dual-task paradigms. If two (or more) tasks undertaken together exceed the available attention capacity, there will be insufficient capacity to optimally perform both tasks and the performance of one or both of the tasks will deteriorate. Impairments in executive function lead to the dual-task paradigm. Dual tasks can be motor-cognitive, cognitive-cognitive, or motor-motor. In a previous study, a negative effect of dual assignment on gait parameters in Type 2 diabetes was observed. It suggests that impaired dual-task capacity in type 2 diabetes may explain the higher incidence of falls in this populationGiven the changes in cognitive function identified in people with poor glycemic control, dual-task testing may provide a functional biomarker for movement impairment and fall risk. A previously published meta-analysis suggested that dual-task testing in people with diabetes better emphasizes deficiencies in functional performance rather than single-task testing, and that dual-task testing can be used to identify people who will start rehabilitation interventions to improve functional performance and reduce the risk of falls. However, although cognitive function declines are common in prediabetic individuals, dual-task performance has not been evaluated and compared with diabetic individuals in previous studies to show the effect of these declines on functional performance. Therefore, the aim of this study is to compare cognitive and motor dual-task performance in individuals with prediabetes and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* be 65 years or older
* Being diagnosed with type 2 diabetes or prediabetes
* Volunteer to participate in the study
* Ability to participate in tests independently
* Getting a score of 24 or higher on the Mini Mental State Test
* Being literate
* Being able to communicate

Exclusion Criteria:

* Cancer patients known to be life-threatening
* Severe respiratory, central, vascular, peripheral and uncontrolled metabolic problems
* Using drugs known to affect the postural control system (eg benzodiazepines)
* Those with peripheral neuropathy
* Those with severe hearing and visual impairments

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Ministry of Health, Karabük Provincial Health Directorate, Barış Family Health Center / 780520 Health Center Safranbolu / Karabük center applied to the center, Dr. Patients over the age of 65 who volunteered to participate in the study, who were followed up by Hasan Hüseyin Mermerkaya, who came on a routine basis, had a blood test within a maximum of 6 months, and were diagnosed with type 2 diabetes or prediabetes, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Timed Get Up and Go Test-Motor and Cognitive Task: | 15 minutes
  The timed up-and-go test is a widely used clinical test to evaluate balance and mobility. The clinical benefit of the test is that it can monitor transitions that require balance control, and mobility skills such as sitting up and walking straight. As the primary task, the participant stands up with the command "Start" from a 46cm standard height chair and walks 3 meters, then turns 180⁰ back and sits on the chair. As a secondary task, he is asked to carry a standardized glass of water without spilling it during the test. As a cognitive task, the participant stands up with the "Start" command from a 46cm standard height chair as the primary task and walks 3 meters, then turns 180⁰ back and sits on the chair. As a secondary task, he is asked to count backwards from 100 by sevens during the test. He will be allowed to practice cognitively in his seat before starting the test. The time elapsed during the test will be recorded.

SECONDARY OUTCOMES:
Short Physical Performance Battery: | 10 minutes
  The Brief Physical Performance Battery is a test used to summarize physical performance based on lower extremity performance, used in populations designated for epidemiological studies of the elderly. It consists of 3 objective tests evaluating lower body function. These; It is a 4 meter walking, standing and standing balance test.
Muscle Strength Measurement | 5 minutes
  Muscle strength will be assessed by hand grip strength for the upper extremity. Individuals' standard grip strength will be measured with a Jamar hand dynamometer (Baseline Evaluation System, New York, USA). The measurement will be made in the test position standardized by the American Association of Hand Therapists, with the patient sitting upright in a chair without arm support, with the shoulder in adduction, the elbow in 90° flexion, the forearm in neutral position, the wrist in 0-30° extension and 0-15° ulnar deviation. While performing the assessment, individuals will be asked to tighten the dynamometer with all their strength and then let it loose completely. This procedure will be repeated in the dominant hand with 1 minute interval between each measurement and the average of these values will be taken in kg/force.
Mini Mental State Test | 10 minutes
  Mini Mental State Test (MMDT) was used in our study for cognitive status assessment. MMDT was first described by Folstein et al. (23) in 1975. The scale was produced as a cognitive assessment tool that can be applied in a short time in the examination of the elderly. The scale has limited specificity for distinguishing clinical syndromes; however, it is a short, useful, valid and standardized method that can be used to evaluate the cognitive level in general.
Fatigue Assessment | 2 minutes
  Fatigue was assessed with the Visual Analog Scale (VAS). VAS, "Are you tired?" It was used to determine the severity of fatigue in elderly individuals who answered yes to the question. VAS is a simple to use, effective, validity and reliability measurement scale (22). In order to determine their fatigue, individuals will be asked to mark the severity of fatigue on a 10 cm scale where the numbers "0" (no fatigue) and "10" (I am unbearably tired) are shown.
Pain Assessment | 2 minutes
  Pain was assessed with the Visual Analogue Scale (VAS). VAS, "Do you have pain?" It was used to determine the severity of pain in elderly individuals who answered yes to the question. VAS is a simple to use, effective, validity and reliability measurement scale (21). Individuals will be asked to mark the severity of pain on a 10 cm scale where the numbers "0" (no pain) and "10" (unbearable pain) are displayed to determine body pain.
Biochemical Analysis | 15 minutes
  The most up-to-date results of blood test results given by individuals within a maximum of 6 months will be recorded by looking at the system. Results of fasting glucose levels, total cholesterol, triglyceride, LDL-cholesterol, HDL-cholesterol, hemoglobin values, urea, creatinine levels of individuals in the research group will be recorded.

REFERENCES:
- [Background] 1. World health Organization (WHO), Diabetes Fact Sheet. Updated October 30th 2018. 2. Zhou B, Lu Y, Hajifathalian K,et al. Worldwide trends in dia- betes since 1980: a pooled analysis of 751 population-based studies with 4.4 million participants. Lancet 2016; 387(10027): .1513-30. 3. Chatterjee S, Peters SAE, Woodward M, Mejia Arango SM, Batty D, Beckett N, et al. Type 2 diabetes as a risk factor for dementia in women compared with men: A pooled analysis of 2.3 million people comprising more than 100,000 cases of dementia. Diabetes Care. 2016. February; 39(2): 300-307. 4. Reyes-García R., Moreno-Pérez Ó., Tejera-Pérez C., Fernández-García D., Bellido-Castañeda V., López de la Torre Casares M., Rozas-Moreno P., Fernández-García J.C., Marco Martínez A., Escalada-San Martín J., et al. A comprehensive approach to type 2 diabetes mellitus-A recommendation document. Endocrinol. Diab. Nutric. 2019;66:443-458. doi: 10.1016/j.endinu.2018.10.010. 5. Schlienger J.-L. Complications du diabète de type 2. Presse Med. 2013;42:839-848. doi: 10.1016/j.lpm.2013.02.313. 6. Diabetes Association of the Republic of China (Taiwan) Executive summary of the DAROC clinical practice guidelines for diabetes care-2018. J. Formos. Med. Assoc. 2019 doi: 10.1016/j.jfma.2019.02.016. 7. Centers for Disease Control and Prevention. National diabetes statistics report: estimates of diabetes and its burden in the United States, 2014. Atlanta: US Department of Health and Human Services; 2014, International Diabetes Federation IDF diabetes atlas 2015. 7th. Brussels: International Diabetes Federation; 2015. 8. Middelbeek RJW, Abrahamson MJ. Diabetes, prediabetes, and glycemic control in the United States: challenges and opportunities. Ann Intern Med. 2014;160:572-573. 9. Forouhi N, Luan J, Hennings S, Wareham N. Incidence of Type 2 diabetes in England and its association with baseline impaired fasting glucose: the Ely study 1990-2000. Diabetic medicine. 2007;24(2):200-7., Nathan DM, Davidson MB, DeFronzo RA, Heine RJ, Henry RR, Pratley R, et al. Impaired fasting glucose and impaired glucose tolerance. Diabetes care. 2007;30(3):753-9. 10. Hu D, Fu P, Xie J, et al. MS for the InterASIA Collaborative Group Increasing prevalence and low awareness, treatment and control of diabetes mellitus among Chinese adults: the InterASIA study. Diabetes Res Clin Pract. 2008;81:250-257. 11. Brannick B, Wynn A, Dagogo-Jack S. Prediabetes as a toxic environment for the initiation of microvascular and macrovascular complications. Exp Biol Med (Maywood) 2016;241:1323-1331. 12. Tuligenga RH, Dugravot A, Tabak AG, et al. Midlife type 2 diabetes and poor glycaemic control as risk factors for cognitive decline in early old age: a post-hoc analysis of the Whitehall II cohort study. Lancet Diabetes Endocrinol. 2014;2:228-235. doi: 10.1016/S2213-8587(13)70192-X. 13. Alosco ML, Gunstad J. The negative effects of obesity and poor glycemic control on cognitive function: a proposed model for possible mechanisms. Curr Diab Rep. 2014. June; 14(6): 495 10.1007/s11892-014-0495. 14. Munshi M, Capelson R, Grande R, Lin S, Hayes M, Milberg W, et al. Cognitive dysfunction is associated with Poor Diabetes Control in Older Adults. Diabetes Care, 2006. August; 29(8): 1794-1799. 10.2337/dc06-0506. 15. Koekkoek PS, Kappelle LJ, van den Berg E, Rutten GE, Biessels GJ. Cognitive function in patients with diabetes mellitus: guidance for daily care. Lancet Neurol. 2015. March; 14(3): 329-340. 10.1016/S1474-4422(14)70249-2. 16. Roriz-Filho S.Sa-Roriz T.M.Rosset I.et al.(Pre)diabetes, brain aging, and cognition.Biochim Biophys Acta. 2009; 1792: 432-443. 17. Woollacott M, Shumway-Cook A. Attention and the control ofposture and gait: a review of an emerging area of research. GaitPosture 2002; 16(1): 1-14. 18. Wollacott M, Shumway-Cook A. Attention and the control of posture and gait; a review of an emerging area of research. Gait Posture 2002; 16: 1- 14. 19. Villafaina S., Collado-Mate D., Domínguez-Muñoz F.J., Fuentes-García J.P., Gusi N. Impact of adding a cognitive task while performing physical fitness tests in women with fibromyalgia: A cross-sectional descriptive study. Medicine (Baltimore) 2018;97:e13791. 20. Omana H, Madou E., Montero-Odasso et all. The Effect of Dual-Task Testing on Balance and Gait Performance in Adults with Type 1 or Type 2 Diabetes Mellitus: A Systematic Review., Current Diabetes ReviewsBentham science Publishers, Current Diabetes Reviews, 2020, Vol.16, no.1-0.